CLINICAL TRIAL: NCT06829589
Title: Assessment of the Retrieval of Economic Incentives and Information Provision on Quality-of-care Indicators for Primary Care Professionals
Brief Title: Retrieval of Economic Incentives and Information on Quality-of-care Indicators in Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Catalan Institute of Health (Other Government)
Responsible Party: Principal Investigator, Josep Vidal-Alaball, MD, PhD, Head of Research, Innovation and Data Analysis, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24/262-P
Record Dates: First submitted 2025-02-05; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Diabetes; Atrium; Fibrillation; Asthma
Keywords: pay-for-performance; primary care; quality-of-care indicators; feedback; healthcare policy; information provision
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Atrial Fibrillation; Asthma

STUDY DESIGN:
Intervention Model Description: Unblinded cluster randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in the Control group will not have any change in their information and incentives schemes.
- Incentive removal (Experimental): Participants will no longer have the economic incentives linked to 7 quality-of-care indicators.
  Interventions: Other: Removal of economic incentives linked to 7 quality-of-care indicators
- Incentive and information removal (Experimental): Participants will no longer have the economic incentives linked to 7 quality-of-care indicators (like in the Incentive removal arm). In addition to this, the information on the indicator results from the online platform for health professionals will be removed.
  Interventions: Other: Removal of economic incentives linked to 7 quality-of-care indicators; Other: Removal of information provision linked to 7 quality-of-care indicators

INTERVENTIONS:
Other: Removal of economic incentives linked to 7 quality-of-care indicators — The 7 intervened indicators will be the following:
  * Blood pressure (BP) control in type-2 diabetes mellitus.
  * BP control in ischemic cardiopathy/cerebrovascular accident.
  * Hypertension: BP control in chronic renal insufficiency.
  * Hypertension: BP control.
  * Diagnostic adequacy of hypertension.
  * Correct treatment of atrial fibrillation.
  * Inhaler verification.
  Professionals randomized to an arm with this intervention will no longer receive an economic reward for reaching a specific goal in the results of these 7 indicators.
  The study guarantees no financial loss since the amount of money linked to these incentives will be automatically given to professionals under the concept of participating in the study.
  Arms: Incentive and information removal; Incentive removal
Other: Removal of information provision linked to 7 quality-of-care indicators — The 7 indicators will be the same as the previous intervention.
  Professionals randomized to an arm with this intervention will no longer see the following in the online platform:
  * Numeric result of the indicator.
  * Color coding to represent indicator result in relation to the yearly goal.
  * 12-month evolution graph.
  Next to the 7 indicator names, only the link to a list of patients that are not fulfilling the indicator criteria will be presented (identifying the patients missing a treatment, a control or any other intervention), since this is considered a tool to support clinical practice beyond informing on the result of an indicator.
  Arms: Incentive and information removal

SUMMARY:
Background: Information provision and economic incentives for professionals are measures aimed at improving quality-of-care in primary care. They are frequently implemented in combination, thus, there is a lack of evidence confirming their individual effectiveness. Since 2006, the Catalan Health Institute (ICS) has implemented a quality improvement system based on a) informing professionals on the result of quality-of-care indicators through an online platform, and simultaneously b) introducing economic incentives in a pay-for-performance (P4P) scheme. There is an unmet need for evidence on the specific impacts of these interventions on quality-of-care.

Aims: Overall, the main aim of the study is to analyze the impact of removing information provision and economic incentives on quality-of-care indicators. Specifically, investigators aim (1) to analyze the effect of removing an economic incentive from a quality-of-care indicator, (2) to analyze the effect of removing information provision from an indicator, (3) to evaluate such effects based on the type of indicator, (4) to evaluate potential spillover effects between indicators linked to the same health problem, and (5) to evaluate potential changes in the professionals' registry patterns.

Methods: The study will be an unblinded cluster randomized clinical trial, with 3 branches: (1) Control, with no changes in the information/incentive schemes; (2) Removal of the economic incentives from a subset of 7 indicators; (3) Removal of the economic incentives and information linked to the 7 indicators. The study duration will be from February to December 2025, with intermediate analyses at 3, 6 and 9 months. The reference population will be the 68 ICS primary care practices (PCPs) in the regions of Catalunya Central, Penedès and Girona. The primary endpoint will be the monthly quality-of-care indicator result of the 7 indicators, and secondary endpoints will include PCP, professional and patient characteristics. The analysis of the intervention effects will be carried out using mixed models and comparing the evolution of results versus the previous years (2019-2024).

DETAILED DESCRIPTION:
Background

Primary care serves as the first point of contact for patients within the healthcare system, addressing key health issues through preventive, curative, and rehabilitative services. Economic incentives, such as pay-for-performance (P4P) schemes, aim to align healthcare professionals' objectives with those of health providers and society by rewarding the achievement of quality-of-care targets. In many cases, P4P is implemented alongside information provision, as seen in the UK's Quality and Outcomes Framework (QOF), where public reporting of quality indicators adds a reputational incentive. However, the interaction between financial and non-financial incentives remains complex, and their long-term effects on quality-of-care continue to be debated.

In Catalonia, the Catalan Institute of Health (ICS) has implemented a quality improvement system since 2006, using the Quality Standard of Care (EQA) framework, which includes 118 evidence-based indicators. This system combines real-time performance feedback through an online platform (information provision) with financial incentives linked to achieving specific targets. While the approach has been well established, many incentivized indicators have plateaued in performance, raising questions about the added value of financial incentives beyond information provision alone in such situations. This study aims to evaluate the impact of removing economic incentives or information on selected EQA indicators, assessing effects by indicator type and exploring interactions between related indicators. The findings will provide crucial insights to optimize incentive strategies and improve healthcare quality in Catalonia.

Aims

General aim: To study the impact of removing economic incentives and/or information provision on quality-of-care indicators among primary care professionals.

Specific aims:

1. To analyze the effect of removing a financial incentive from an indicator: to provide evidence on what happens when points from a quality-of-care indicator linked to the Catalan Health Institute's (ICS) Direcció per Objectius (DPO) are removed, meaning that a specific indicator or a set of indicators for a clinical condition is no longer financially incentivized.
2. To analyze the effect of partially removing information from an indicator: to assess the additional impact of withdrawing part of the information related to a specific indicator or a set of indicators for a particular condition.
3. To analyze the effects of objectives 1 and 2 based on indicator type: to evaluate whether the observed effects differ according to certain characteristics of the indicators: (a) indicators that have had consistently high results for years (plateaued) and have high clinical relevance; (b) indicators primarily related to data recording; (c) sets of indicators associated with a specific condition.
4. To assess potential spillover effects on other indicators: to determine whether removing incentives and/or information from an indicator affects other indicators related to the same clinical condition that remain incentivized and publicly reported.
5. To evaluate changes in professionals' recording patterns: to determine whether the presence or absence of financial incentives for indicators leads to changes in the way healthcare professionals record data.

Study design

A cluster-randomized clinical trial without blinding. The study will include the following groups (further detail provided in the Arms and Interventions section):

* Control Group: No changes in the information and incentive scheme.
* Intervention 1: Removal of the financial incentive for a selected set of indicators.
* Intervention 2: Removal of the same financial incentives as in Intervention 1, along with the removal of related information in the online platform for professionals (numeric result of the indicator, 12-month evolution lineplot, number of patients not fulfilling the indicator criteria, degree of accomplishment of the indicator in relation to specific goals using a traffic light color coding)

Study Period and Duration

The study will take place from February 2025 to December 2025. Weekly monitoring of the primary outcome variable will be conducted, with interim analyses at 3, 6, and 9 months.

Setting and Target Population

The study will be conducted in primary care practices (PCPs) of the Catalan Health Institute (ICS). To minimize interference from territorial management incentives and encourage participation, the trial will be carried out in three regional health management areas: Catalunya Central, Penedès and Girona. These regions were selected after discussions with their management teams and agreement on the study's implementation.

The trial will be conducted at the level of individual healthcare professionals (family physicians and nurses). However, randomization will be performed at the PCP level, ensuring that all professionals within the same PCP are assigned to the same arm of the study.

Statistical analysis

The analysis will be conducted at both the individual professional and EAP levels and will include all professionals from both intervention and control EAPs, regardless of whether they have used clinical decision support tools (SISAP web and/or patient lists). The analysis will follow an intention-to-treat (ITT) approach.

First, a descriptive analysis will be performed to assess the characteristics of each group, ensuring balance across different EAP and professional-level characteristics. Balance will be evaluated using the standardized mean difference (SMD), where an SMD > 0.1 will indicate imbalance.

The primary analysis will be focused on the effect of incentive and information withdrawal. The effect of removing financial incentives and removing both incentives and information will be analyzed using mixed-effects models, which account for intra-cluster variability and EAP-level clustering effects. A linear mixed-effects model will be used, considering both fixed and random effects. Fixed effects will include the intervention and any imbalanced covariates (based on SMD > 0.1). Random effects will account for variability within clusters (EAPs). Results will be reported as effect estimates with 95% confidence intervals (CI95%). In addition to the above, pre-post models will also be conducted to compare current vs. past performance for the same indicators.These analyses will be conducted at 3, 6, 9, and 12 months.

To assess for changes in documentation patterns (objective #5), the study will compare the distribution of systolic (SBP) and diastolic blood pressure (DBP) values recorded for patients included in blood pressure-related indicators across control and intervention groups. The descriptive statistics mean ± standard deviation (SD) and median ± interquartile range (IQR) will be reported. T-tests will be used to compare mean differences between groups.

ANOVA followed by Tukey's post-hoc test will be used for multiple comparisons. If normality or homoscedasticity assumptions are violated, non-parametric tests will be applied instead. Statistical significance (α = 0.05) will be adjusted for multiple comparisons to control for Type I errors.

Informed consent

The regional and PCP management teams have the authority to decide which indicators contribute to the P4P scheme for each professional. This system allows a certain flexibility in awarding economic incentives for professionals. Given this framework, individual informed consent from professionals is not deemed necessary. However, the study will be presented to the directors of the participating PCPs and their agreement to participate in the study will be collected with study participation acceptance forms. These stakeholders will be fully informed about the study, including the fact that their professionals will be enrolled in a randomized clinical trial, and that professionals in the intervention groups (where some indicators have their points removed) will not experience any financial penalty. As a secondary validation, professionals will implicitly confirm their consent when signing their P4P scheme agreements. If any professional disagrees with their P4P scheme, they will be excluded from the study, and no intervention will be applied to them.

ELIGIBILITY:
Inclusion Criteria:

* Any general practitioner or nurse working in a primary care practice.
* Having enough clinical activity to be included in the pay-for-performance schemes by the PCP director.
* Belonging to a PCP in the regions of Catalunya Central, Penedès or Girona.
* Belonging to a PCP whose director accepted to participate in the study.

Exclusion Criteria:

* PCPs with very low overall quality-of-care scores (<60%).
* Professionals who did not sign the pay-for-performance contracts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1614 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Monthly percentage of achievement of the 7 quality-of-care indicators | Evaluation will be carried out at baseline and at months 3, 6, 9 and 12 of the year
  The result of the quality-of-care indicators is calculated as the % of achievement. This is routinely computed by the Catalan Health Institute Information Systems using the electronic health records.

OTHER OUTCOMES:
Monthly percentage of achievement stratified by practice rurality | Baseline and at 1 year
  Urban primary care practices (PCPs) are considered those in municipalities with >10,000 inhabitants and a population density >150 people/km2. The rest are considered rural PCPs.
Monthly percentage of achievement stratified by social deprivation index | Baseline and at 1 year
  The social deprivation index built to assign the budgets of the PCPs in Catalonia will be used (PMID: 30595339).
Monthly percentage of achievement stratified by PCP accessibility | Baseline and at 1 year
  Accessibility will be defined as the probability of patients to be visited by the GP or nurse in 48 hours. It will be a monthly measure.
Monthly percentage of achievement stratified by PCP frequentation | Baseline and at 1 year
  Frequentation will be defined as the average annual attendance time per patient in the PCP.
Monthly percentage of achievement stratified by sex of the professional | Baseline and at 1 year
  Male and female professionals.
Monthly percentage of achievement stratified by specialty of the professional | Baseline and at 1 year
  General practitioners and nurses.
Monthly percentage of achievement stratified by age of the professional | Baseline and at 1 year
  5-year age intervals will be considered.
Monthly percentage of achievement stratified by years worked | Baseline and at 1 year
  Years worked in the Catalan Health Institute.
Monthly percentage of achievement stratified by sex distribution in the patient panels | Baseline and at 1 year
  % of male and female patients in the panel.
Monthly percentage of achievement stratified by % of immigrant population in the patient panels | Baseline and at 1 year
  % of people with a non-Spanish nationality in the patient panel.

CONTACTS AND LOCATIONS:
Locations (68):
- Spain (68):
  - ABS Artés, Artés, Barcelona
  - ABS Berga, Berga, Barcelona
  - ABS Calaf, Calaf, Barcelona
  - ABS Canet de Mar, Canet de Mar, Barcelona
  - ABS Capellades, Capellades, Barcelona
  - ABS Cardona, Cardona, Barcelona
  - ABS Moià, Castellterçol, Barcelona
  - ABS Cubelles-Cunit, Cubelles, Barcelona
  - EAP Penedès Rural Est, Els Monjos, Barcelona
  - EAP Penedès Rural Oest, Els Monjos, Barcelona
  - ABS Baix Berguedà, Gironella, Barcelona
  - ABS Alt Berguedà, Guardiola de Berguedà, Barcelona
  - ABS Igualada urbana, Igualada, Barcelona
  - ABS Anoia Rural, La Pobla de Claramunt, Barcelona
  - ABS Manlleu, Manlleu, Barcelona
  - ABS Manresa-2, Manresa, Barcelona
  - ABS Manresa-4, Manresa, Barcelona
  - ABS Montserrat, Monistrol de Montserrat, Barcelona
  - ABS Navàs/Balsareny, Navàs, Barcelona
  - ABS Piera, Piera, Barcelona
  - ABS Pineda de Mar, Pineda de Mar, Barcelona
  - ABS Lluçanès, Prats de Lluçanès, Barcelona
  - EAP Roda de Ter, Roda de Ter, Barcelona
  - ABS Sallent, Sallent, Barcelona
  - ABS Navarcles - Sant Fruitós de Bages, Sant Fruitós de Bages, Barcelona
  - ABS Sant Hipòlit de Voltregà, Sant Hipòlit de Voltregà, Barcelona
  - ABS Sant Joan de Vilatorrada, Sant Joan de Vilatorrada, Barcelona
  - EAP Ribes-Olivella, Sant Pere de Ribes, Barcelona
  - EAP Roquetes-Canyelles, Sant Pere de Ribes, Barcelona
  - ABS Sant Quirze de Besora, Sant Quirze de Besora, Barcelona
  - ABS Sant Sadurní d'Anoia, Sant Sadurní d'Anoia, Barcelona
  - ABS Sant Vicenç de Castellet, Sant Vicenç de Castellet, Barcelona
  - ABS Santa Eugènia de Berga, Santa Eugènia de Berga, Barcelona
  - ABS Santa Margarida de Montbui, Santa Margarida de Montbui, Barcelona
  - ABS Santpedor, Santpedor, Barcelona
  - ABS Sitges, Sitges, Barcelona
  - ABS Súria, Súria, Barcelona
  - ABS Tona, Tona, Barcelona
  - ABS Tordera, Tordera, Barcelona
  - ABS La Vall de Ges, Torelló, Barcelona
  - ABS Vic-1 Nord, Vic, Barcelona
  - EAP Vilafranca del Penedès-1, Vilafranca del Penedès, Barcelona
  - EAP Vilafranca del Penedès-2, Vilafranca del Penedès, Barcelona
  - ABS Vilanova del Camí, Vilanova del Camí, Barcelona
  - ABS Vilanova i la Geltrú-1, Vilanova i la Geltrú, Barcelona
  - ABS Vilanova i la Geltrú-2, Vilanova i la Geltrú, Barcelona
  - ABS Arbúcies/Sant Hilari, Arbúcies, Girona
  - EAP Bàscara, Bàscara, Girona
  - ABS Besalú, Besalú, Girona
  - ABS Camprodon, Camprodon, Girona
  - ABS Celrà, Celrà, Girona
  - ABS Figueres, Figueres, Girona
  - ABS La Jonquera, la Jonquera, Girona
  - ABS Llançà, Llançà, Girona
  - ABS Olot, Olot, Girona
  - ABS Ripoll, Ripoll, Girona
  - ABS Roses, Roses, Girona
  - ABS Salt, Salt, Girona
  - ABS Sant Feliu de Guíxols, Sant Feliu de Guíxols, Girona
  - ABS Santa Coloma de Farners, Santa Coloma de Farners, Girona
  - ABS Sarrià de Ter, Sarrià de Ter, Girona
  - ABS Sils-Vidreres-Maçanet de la Selva, Sils, Girona
  - EAP Vilafant, Vilafant, Girona
  - ABS Santa Coloma de Queralt, Santa Coloma de Queralt, Tarragona
  - ABS Girona-1, Girona
  - ABS Girona-3, Girona
  - ABS Girona-2, Girona
  - ABS Girona-4, Girona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roland M, Guthrie B. Quality and Outcomes Framework: what have we learnt? BMJ. 2016 Aug 4;354:i4060. doi: 10.1136/bmj.i4060. PMID 27492602
- [Background] Roland M, Dudley RA. How Financial and Reputational Incentives Can Be Used to Improve Medical Care. Health Serv Res. 2015 Dec;50 Suppl 2(Suppl 2):2090-115. doi: 10.1111/1475-6773.12419. Epub 2015 Nov 17. PMID 26573887
- [Background] Allen T, Whittaker W, Kontopantelis E, Sutton M. Influence of financial and reputational incentives on primary care performance: a longitudinal study. Br J Gen Pract. 2018 Dec;68(677):e811-e818. doi: 10.3399/bjgp18X699797. Epub 2018 Nov 5. PMID 30397016
- [Background] Eijkenaar F, Emmert M, Scheppach M, Schoffski O. Effects of pay for performance in health care: a systematic review of systematic reviews. Health Policy. 2013 May;110(2-3):115-30. doi: 10.1016/j.healthpol.2013.01.008. Epub 2013 Feb 4. PMID 23380190
- [Background] Roland M, Campbell S. Successes and failures of pay for performance in the United Kingdom. N Engl J Med. 2014 May 15;370(20):1944-9. doi: 10.1056/NEJMhpr1316051. No abstract available. PMID 24827040
- [Background] Wagenschieber E, Blunck D. Impact of reimbursement systems on patient care - a systematic review of systematic reviews. Health Econ Rev. 2024 Mar 16;14(1):22. doi: 10.1186/s13561-024-00487-6. PMID 38492098
- [Background] Mendelson A, Kondo K, Damberg C, Low A, Motuapuaka M, Freeman M, O'Neil M, Relevo R, Kansagara D. The Effects of Pay-for-Performance Programs on Health, Health Care Use, and Processes of Care: A Systematic Review. Ann Intern Med. 2017 Mar 7;166(5):341-353. doi: 10.7326/M16-1881. Epub 2017 Jan 10. PMID 28114600
- [Background] Zaresani A, Scott A. Is the evidence on the effectiveness of pay for performance schemes in healthcare changing? Evidence from a meta-regression analysis. BMC Health Serv Res. 2021 Feb 24;21(1):175. doi: 10.1186/s12913-021-06118-8. PMID 33627112
- [Background] Chauhan BF, Jeyaraman MM, Mann AS, Lys J, Skidmore B, Sibley KM, Abou-Setta AM, Zarychanski R. Behavior change interventions and policies influencing primary healthcare professionals' practice-an overview of reviews. Implement Sci. 2017 Jan 5;12(1):3. doi: 10.1186/s13012-016-0538-8. PMID 28057024
- [Background] Coma E, Ferran M, Mendez L, Iglesias B, Fina F, Medina M. Creation of a synthetic indicator of quality of care as a clinical management standard in primary care. Springerplus. 2013 Dec;2(1):51. doi: 10.1186/2193-1801-2-51. Epub 2013 Feb 13. PMID 23450738